CLINICAL TRIAL: NCT01283607
Title: Treatment of Depression and Anxiety by an E-health Cognitive Behavioral Therapy (Digicoach) in Women Treated by in Vitro Fertilization (IVF)
Brief Title: E-health Cognitive Behavioral Therapy in Women Treated by in Vitro Fertilization (IVF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Nijmegen (Other)
Collaborators: Stichting Nuts Ohra (Other)
Responsible Party: Principal Investigator, Angelique van Dongen, MD, University Medical Center Nijmegen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Digicoach
Record Dates: First submitted 2011-01-21; First posted 2011-01-26 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-11

CONDITIONS: Depression; Anxiety; Infertility
Keywords: in vitro fertilization; e-health; cognitive behavioral therapy; psychosocial risk profile; emotional maladjustment
MeSH Terms: conditions — Depression; Anxiety Disorders; Infertility

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Digicoach (Active Comparator): Women randomized in the Digicoach group will be treated by the Digicoach therapy. Digicoach is an e-health cognitive behavioral therapy with 4-12 weekly sessions especially developed for in vitro fertilization (IVF) women. Digicoach is facilitated by an e-therapist. The investment for the weekly home work assignments is about one and a half hour. Digicoach consist of different modules (e.g. stress reduction, acceptance). Digicoach starts before the hormonal down regulation as the start of the IVF procedure and ends three weeks after the pregnancy test.
  Interventions: Behavioral: Digicoach
- Control (No Intervention): Women in the control group will get the usual treatment, there will be no additional intervention.

INTERVENTIONS:
Behavioral: Digicoach — Digicoach is an e-health cognitive behavioral therapy with 4-12 weekly sessions especially developed for IVF women. Digicoach is facilitated by an e-therapist. The investment for the weekly home work assignments is about one and a half hour. Digicoach consist of different modules (e.g. stress reduction, acceptance). Digicoach starts before the hormonal down regulation as the start of the IVF procedure and ends three weeks after the pregnancy test.
  Arms: Digicoach

SUMMARY:
Yearly, 15,000 Dutch in vitro fertilization (IVF) cycles are performed for subfertility with a pregnancy rate of 26%. A failed cycle has great emotional impact; 20-25% of the women has relevant forms of depression/anxiety even after 6 months. For such maladjustment a risk profile has been identified and translated into a screening tool. Identification of women at risk enables a timely and tailored (individual's needs) cognitive behavioral therapy (CBT), which reduces more serious maladjustment and corresponding costs.

Aim: To investigate the effectiveness of an e-health CBT (digital coaching, Digicoach) in women ongoing IVF and having been screened at risk.

Design: A single-centered randomised controlled trial comparing Digicoach (intervention) with standard care (control).

Digicoach: an e-health CBT with 4-12 weekly sessions starting before an IVF cycle, following a woman's IVF course and covering in modules the main problems: depressed mood, anxiety, strong focus on child wish and acceptance.

Main outcome measures: anxiety and depression occurrence rate 3 weeks after an unsuccessful IVF cycle. Secondary outcome measures: 1. (para)medical consumption, 2. quality of life, 3. productivity loss and 4. IVF outcome. Data are collected by questionnaires, diaries, medical record audit and page view registrations.

Process evaluation: Individual's use (e.g. module progress, completion rate), experiences, (e.g. satisfaction and usability) and potential barriers for implementation are evaluated.

Economic evaluation: studied during the Digicoach exposures from a societal perspective. Incremental costs (costs/%avoidance of depression/anxiety) are determined by comparing both study groups.

Power/data analysis: To detect a 29% difference in the depression/anxiety occurrence rates (alfa=0.05 and beta=0.80) 58 unpregnant IVF women are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* women screened as 'at risk' for emotional maladjustment after In vitro fertilization (IVF) by a screening tool

Exclusion Criteria:

* impossibility to use Internet
* impossibility to write or read the Dutch language
* high screening scores requiring immediate intervention

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2011-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
scores on anxiety and depression | three months after an in vitro fertilization (IVF) cycle.
  anxiety and depression rates three weeks after an unsuccessful IVF cycle, scored by the Hospitality Anxiety Depression Scale (HADS), we also measure the scores during the IVF cycle and three months after the IVF cycle.

SECONDARY OUTCOMES:
(para)medical consumption | during the IVF cycle
  by questionnaires
process evaluation of the webbased cognitive behavioral therapy (CBT) | after the IVF cycle
  process evaluation will be investigated by the individual's use of Digicoach (page view registration) and the patients' and professionals' experiences with Digicoach (questionnaires).
productivity loss | during the IVF cycle
  by questionnaires
health related quality of life | before, during, three weeks and three months after the IVF cycle
  by questionnaire using FertiQol (Fertility Quality of Life questionnaire), a validated screening instrument measuring quality of life related to fertility treatment
IVF outcome | three weeks after the IVF cycle
  by questionnaire and medical record viewing
economical evaluation | three months after the IVF cycle
  cost effectiveness of the e-health cognitive behavioral therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jan A Kremer, Ph.D. M.D., Study Director — Radboud University Medical Center; Chris M Verhaak, Ph.D., Study Chair — Radboud University Medical Center; Willianne L Nelen, Ph.D. M.D., Study Chair — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, department of obstetrics and gynecology, Nijmegen, Nijmegen, Netherlands

REFERENCES:
- [Background] Verhaak CM, Smeenk JM, van Minnen A, Kremer JA, Kraaimaat FW. A longitudinal, prospective study on emotional adjustment before, during and after consecutive fertility treatment cycles. Hum Reprod. 2005 Aug;20(8):2253-60. doi: 10.1093/humrep/dei015. Epub 2005 Apr 7. PMID 15817584
- [Background] Verhaak CM, Lintsen AM, Evers AW, Braat DD. Who is at risk of emotional problems and how do you know? Screening of women going for IVF treatment. Hum Reprod. 2010 May;25(5):1234-40. doi: 10.1093/humrep/deq054. Epub 2010 Mar 13. PMID 20228392
- [Derived] van Dongen AJ, Nelen WL, IntHout J, Kremer JA, Verhaak CM. e-Therapy to reduce emotional distress in women undergoing assisted reproductive technology (ART): a feasibility randomized controlled trial. Hum Reprod. 2016 May;31(5):1046-57. doi: 10.1093/humrep/dew040. Epub 2016 Mar 10. PMID 26965429